CLINICAL TRIAL: NCT00913549
Title: Bioequivalency Study of Dosage Forms of Clemastine 2.68 mg Tablets
Brief Title: To Demonstrate the Relative Bioequivalency Study of Dosage Forms of Clemastine 2.68 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 239-04
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-06

CONDITIONS: Allergy
Keywords: Antihistamine
MeSH Terms: conditions — Hypersensitivity | interventions — Clemastine

ARMS (2):
- 1 (Experimental): Clemastine Fumarate Tablets, 2.68 mg (Cord Laboratories)
  Interventions: Drug: Clemastine Fumarate Tablets, 2.68 mg (Cord Laboratories)
- 2 (Experimental): Tavist Tablets, 2.68 mg (Sandoz Pharmaceutical Corp.)
  Interventions: Drug: Tavist Tablets, 2.68 mg (Sandoz Pharmaceutical Corp.)

INTERVENTIONS:
Drug: Clemastine Fumarate Tablets, 2.68 mg (Cord Laboratories)
  Arms: 1
Drug: Tavist Tablets, 2.68 mg (Sandoz Pharmaceutical Corp.)
  Arms: 2

SUMMARY:
To demonstrate the relative bioequivalency study of dosage forms of Clemastine 2.68 mg tablets.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 1989-12; Primary Completion 1990-01 (Actual); Study Completion 1990-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 19 days

CONTACTS AND LOCATIONS:
Overall Officials: James C. Kisicki, M.D., Principal Investigator — Harris Laboratories, Incorporated